CLINICAL TRIAL: NCT02433574
Title: Phase I Study: Locally Invasive NSCLC Treated With NEo-Adjuvant Stereotactic Body Radiotherapy and REsection
Brief Title: Locally Invasive NSCLC Treated With NEo-Adjuvant Stereotactic Body RadioTherapy and REsection
Acronym: LINNEARRE-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juravinski Cancer Center (Other)
Responsible Party: Principal Investigator, Theo Tsakiridis, M.D., Ph.D., FRCPC, Radiation Oncologist, Associate Professor, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LINNEARRE-I
Record Dates: First submitted 2015-02-04; First posted 2015-05-05 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Non-Small-Cell Lung Cancer; Carcinoma
Keywords: radiosurgery; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant stereotactic body radiation (Experimental): Single arm study. Four cohorts of 5 patients will undergo neo-adjuvant SBRT for lung cancer. Eligible patients will have operable, borderline resectable lung cancer , they will be treated with SBRT, prior to undergoing surgical resection.
  Interventions: Radiation: Neoadjuvant Stereotactic body radiation (SBRT)

INTERVENTIONS:
Radiation: Neoadjuvant Stereotactic body radiation (SBRT) — Dose escalation of neo-adjuvant SBRT in operable patients with locally advanced non-small cell lung cancer.
  The first cohort will be treated with a dose of 35 Gy in 10 fractions, the second cohort will be treated with a dose of 40 Gy in 10 fractions, the third cohort will be treated with a dose of 45 Gy in 10 fractions, the fourth cohort will be treated with a dose of 50 Gy in 10 fractions. The SBRT doses will be escalated only once all patients in the previous cohort will have completed safely their treatments.

SUMMARY:
Despite improved staging and operative techniques, the rate of incomplete resection (R1) of NSCLC has remained significant over the last decades. Patients with R1 resection have significantly worse survival compared to those with complete resection (R0).

This is a phase I study that investigates the feasibility and safety of delivering Stereotactic Body Radiotherapy (SBRT) to patients with locally invasive NSCLC (cT3-4, N0-1) who are at risk for incomplete resection.

Twenty patients with NSCLC will be treated with SBRT followed by surgery and appropriate adjuvant therapy. Patients will be divided into groups, of 5 patients each, treated with escalating doses (35, 40, 45 and 50 Gy) in 10 daily fractions.

The primary outcome is the feasibility i.e. the ability to complete safely SBRT and surgery (within 6 weeks). Secondary outcomes include acute and late adverse events, R0/R1/R2 rates and secondary surrogates of feasibility.

If successful, this study will lead to further evaluation of pre-operative SBRT in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are aged 18 years or older,
* with biopsy proven NSCLC,
* clinically staged T3-T4 marginally resectable i.e. deemed at risk to achieve <R0 resection (such as invasion of critical mediastinal or hilar structures, nodal extra-capsular extension, chest wall, vertebral bodies, compromised bronchial stump margin, based on CT images of the chest).
* Patients also need to be pathologically staged N0-1 disease,
* with an SBRT CTV≤200cm3, based on planning CT images.
* ECOG status is required to be <2 within 4 weeks prior to registration and
* patients must be deemed medically operable by the surgical team.

Exclusion Criteria:

* Patients will be excluded if they are deemed medically inoperable by the surgical team
* and have a weight loss of ≥10% within 3 months prior to pathological diagnosis.
* Patients will also have no absolute contraindication to RT such as connective tissue disease, pacemaker-dependent patient with the pacemaker receiving higher than tolerance dose, had no had previous RT to the current region of the study, that would result in overlap of RT fields,
* patients must have no plans to receive other local therapy while on study, except at disease progression,
* patients have not had other malignancy within 2 years prior to the study (other than non-melanomatous skin cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of SBRT followed by surgery (proportion of patients who can undergo 10 fractions of SBRT followed by Surgery) | 18 months
  Feasibility of neo-adjuvant SBRT followed by surgery. This will be measured as the proportion of patients who can undergo 10 fractions of SBRT followed by Surgery as scheduled (within 6 weeks from registration).

SECONDARY OUTCOMES:
Early safety of SBRT-S through collection of serious adverse events (CTCAE version 4.0 grade 3 or higher) from beginning of SBRT to 4 weeks after completion of surgery. | 18 months
Late safety profile of SBRT-S through collection of surgical complication rates assessed at 6 and 18 months post-registration (thus 30 months from opening of the study, assuming it takes 1 year to complete accrual). | 30 months
  Complications recorded include incidence of bronchopleural fistula, esophageal fistula, wound healing complications (dehiscence, infection) and post-operative pulmonary complications).
Secondary feasibility outcomes (including accrual rate, consent rate, rates of deviation from scheduled treatment plan, and reasons for delay) | 18 months
  These include accrual rate, consent rate, rates of deviation from scheduled treatment plan of 6 weeks, and reasons for delay)
Pathological response following neoadjuvant SBRT (proportion of R0, R1 and R2 resections) | 18 months
  To determine the proportion of R0, R1 and R2 resections after neoadjuvant SBRT.
Pathologic changes associated with neo-adjuvant SBRT with analysis of irradiated tissues | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Tsakiridis, M.D., Ph.D., Principal Investigator — Juravinski Cancer Center
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Nguyen NA, Isfahanian N, Pond G, Hanna W, Cutz JC, Wright J, Swaminath A, Shargall Y, Chow T, Wierzbicki M, Okawara G, Quan K, Finley C, Juergens R, Tsakiridis T. A Novel Neoadjuvant Therapy for Operable Locally Invasive Non-Small-Cell Lung Cancer. Phase I Study of Neoadjuvant Stereotactic Body Radiotherapy. LINNEARRE I (NCT02433574). Clin Lung Cancer. 2017 Jul;18(4):436-440.e1. doi: 10.1016/j.cllc.2017.01.007. Epub 2017 Jan 31. PMID 28215851